CLINICAL TRIAL: NCT06626620
Title: Randomized Controlled Trial of Intravenous Magnesium Sulfate Versus Terbutaline for Children in the Management of Acute Exacerbation of Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Collaborators: Nishtar Medical University (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NISHTARASTHMASTUDY
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Exacerbation of Asthma
Keywords: Asthma; intravenous; magnesium sulfate; terbutaline
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Magnesium Sulfate (Experimental): Magnesium sulfate, a smooth muscle relaxant, has been shown to have bronchodilatory effects by inhibiting calcium influx into smooth muscle cells.
  Interventions: Drug: Magnesium Sulphate infusion
- IV Terbutaline (Experimental): Terbutaline, a beta-2 agonist, is used intravenously to provide systemic bronchodilation when inhaled bronchodilators are not effective.
  Interventions: Drug: Terbutaline Infusion

INTERVENTIONS:
Drug: Magnesium Sulphate infusion — Received IV magnesium sulfate (50 mg/kg up to a maximum dose of 2 g) administered over 20 minutes
  Other Names: IV MgSO4
  Arms: IV Magnesium Sulfate
Drug: Terbutaline Infusion — Received IV terbutaline (10 mcg/kg bolus followed by a continuous infusion of 0.4 mcg/kg/min) for up to 4 hours
  Arms: IV Terbutaline

SUMMARY:
This study aimed to fill this gap by comparing the effectiveness of intravenous magnesium sulfate versus terbutaline in children with acute asthma exacerbations, providing evidence-based guidance for clinicians in emergency settings.

DETAILED DESCRIPTION:
Despite the established roles of both magnesium sulfate and terbutaline in the management of severe asthma exacerbations, there is limited comparative data on their efficacy and safety in the pediatric population. Understanding the relative benefits and risks of these therapies is crucial for optimizing treatment strategies and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Known cases of asthma
* Minimum duration of asthma as 6 months
* Presenting with acute exacerbation of asthma
* Requiring emergency treatment.

Exclusion Criteria:

* Children having chronic respiratory diseases (cystic fibrosis, bronchopuonary dysplasia)
* Children with cardiac diseases
* Children who were hospitalized in the past 2-weeks due to any reasons
* Children using oral or intravenous corticosteroids or other systemic medications
* Children who were unable to undergo PEFR measurements due to any reasons

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Post-treatment PEFR | 4 hours
  Post-treatment, children response to treatment was measured by noting PEFR

SECONDARY OUTCOMES:
Oxygen Saturation | 4 hours
  Post-treatment, oxygen saturation was measured using Spirometry
Heart Rate | 4-hours
  Post-treatment, heart rate was measured
Respiratory rate | 4 hours
  Post-treatment, heart rate was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Zulqarnain, FCPS, Study Director — Department of Pediatrics, Nishtar Hospital, Multan, Pakistan; Muhammad Salman, FCPS, Principal Investigator — Department of Pediatrics, Nishtar Hospital, Multan
Locations (1):
- Nishtar Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No